CLINICAL TRIAL: NCT07247539
Title: Diyalizat Saf Su Dijital Takip Sistemi
Brief Title: Preventing Hemolysis and Reducing Reverse Osmosis Waste With Instantaneous Measurement of Water Quality and Early Warning System in Hemodialysis: A New Method, "Pure Water Eye"
Acronym: HEMOWAQNEWS
Status: Completed | Type: Observational
Sponsor: Usak State Hospital (Other)
Responsible Party: Principal Investigator, Ender Hur, Professor, Usak State Hospital
Other Study IDs: 699-699-03
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Water Quality; Water Consumption; Water-Related Diseases; Hemodialysis Complication
MeSH Terms: conditions — Waterborne Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: Pure Water Eye Continuous Monitoring System — Pure Water Eye Continuous Monitoring System (Continuous measurement of pH, conductivity, chlorine, turbidity, and TDS)

SUMMARY:
This study validates a novel, continuous, and instantaneous water quality monitoring method, the "Pure Water Eye," for hemodialysis (HD) systems. Current periodic testing leaves patients vulnerable to acute, severe complications like hemolysis due to sudden, undetectable failures in water quality (e.g., chlorine spikes, pH changes). The "Pure Water Eye" system continuously monitors five key parameters to establish an early warning mechanism, significantly increasing patient safety and allowing for the safe optimization of Reverse Osmosis (RO) water usage, thereby reducing water waste. This system is the first of its kind in Turkey, and globally, it addresses a critical gap where instantaneous and continuous monitoring of HD water quality is not standard practice.

DETAILED DESCRIPTION:
The safety of hemodialysis is critically dependent on the quality of the water used, as large volumes directly contact the patient's blood. The current standard of relying on periodic measurements (daily or weekly) fails to detect instantaneous fluctuations in contaminants (e.g., pH, conductivity, chlorine), which can lead to catastrophic events like hemolysis. The "Pure Water Eye" system was developed to perform four measurements per minute across five key parameters: pH, conductivity, chlorine, turbidity, and TDS. This prospective observational study investigated three scenarios: 1) Standard RO measurement, 2) RO waste water reduced by 50%, and 3) RO waste water directly routed back to the raw water tank. The study successfully demonstrated that continuous monitoring is vital for detecting sudden risk moments and is the only safe method for optimizing RO waste reduction without compromising water safety.

ELIGIBILITY:
Inclusion Criteria: Hemodialysis Centre -

Exclusion Criteria:None

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Usak Education and Research Hospital Hemodialysis Centre
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of water quality parameters (pH, Chlorine, Conductivity) exceeding safe Hemodialysis guidelines limits as detected by the Pure Water Eye's instantaneous monitoring system, demonstrating the failure rate missed by standard periodic testing. | through study completion, an average of 3 months
Comparison of water conservation efficiency (reduction in RO waste water volume) between standard RO procedures and the optimized RO waste reduction scenario (Scenario 2: 50% waste reduction) safely managed by instantaneous monitoring. | through study completion, an average of 3 months

SECONDARY OUTCOMES:
Validation of the correlation between instantaneous conductivity measurements and TDS (Total Dissolved Solids) readings to confirm the accuracy of the new method's core functionality. | through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Usak Education and Research Hospital, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] de Oliveira RM, de los Santos CA, Antonello I, d'Avila D. Warning: an anemia outbreak due to chloramine exposure in a clean hemodialysis unit--an issue to be revisited. Ren Fail. 2009;31(1):81-3. doi: 10.1080/08860220802546503. PMID 19142815
- [Result] Kasparek T, Rodriguez OE. What Medical Directors Need to Know about Dialysis Facility Water Management. Clin J Am Soc Nephrol. 2015 Jun 5;10(6):1061-71. doi: 10.2215/CJN.11851214. Epub 2015 May 15. PMID 25979976
- [Result] Barraclough KA, Moller S, Blair S, Knight R, Agar JW, McAlister S, White A, Sypek M. Updating the Data: The Resource Consumption of Modern-Day Hemodialysis Systems. Kidney Int Rep. 2024 Feb 12;9(5):1521-1524. doi: 10.1016/j.ekir.2024.02.010. eCollection 2024 May. No abstract available. PMID 38707837